CLINICAL TRIAL: NCT00169637
Title: Evaluation of the Efficacy and Safety of Recombinant Human Growth Hormone (rhGH) in the Treatment of Children With Short Bowel Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Alain Lachaux, Hospices Civils de Lyon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2002.301
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2008-10-31 (Estimated); Status verified 2008-06

CONDITIONS: Short Bowel Syndrome
Keywords: Short bowel syndrome; Growth hormone; Children
MeSH Terms: conditions — Short Bowel Syndrome

INTERVENTIONS:
Drug: rhGH

SUMMARY:
This is a randomized controlled, parallel group, open label versus "no treatment" trial which evaluate the efficacy of rhGH on weaning off parenteral nutrition in children with short bowel syndrome.The total follow-up is 14 months; 4 months for each group after randomization; At the end of the first four months: the treated group will be followed within 6 months, the untreated group will receive compassionately rhGH for 4 months and followed-up for 6 months after the end of the treatment period.

ELIGIBILITY:
Inclusion Criteria:

Age 3-18 year with a bone age test under 18-year Children with short bowel syndrome and intestinal insufficiency, the remaining bowel length should be under 80 cm after the first post-surgical period.

Parenteral nutrition dependency: under parenteral nutrition for at least 3 years with parenteral glycolipidic diet > or = 30% of the total caloric need for age. The parenteral diet should have been stable for at least 3 months.

Parents consent

Exclusion Criteria:

Over 20% change in caloric daily requirement within the last 6 months before inclusion.

Surgery on digestive tube within the last 3 months. Administration of drugs targeting digestion (decontamination, macrobiotic, gastric dressing, chelating agents of biliary salts) within the last month.

History or presence of tumoral process, leukaemia, minor intracranial hypertension, epiphysiolysis, carpal tunnel syndrome.

Ongoing infection (fever and inflammatory biologic syndrome), progressive inflammatory syndrome.

Heart failure, renal and respiratory insufficiency. Allergy to solvent. Any condition making impossible the follow-up of the patient during the study. Person participating in another clinical trial or taking another medication under investigation within one month before inclusion.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2006-06; Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of rhGH compared to "no treatment" on partial or total weaning off of parenteral nutrition in children with short bowel syndrome after 4 months

SECONDARY OUTCOMES:
Evaluate the persistent efficacy (remaining rate of weaning off) 6 months after rhGH discontinuation.
To evaluate the intestinal absorption (input-output within 3 days) at the end of the randomized study (month 4) and at the end of study (month 14)
To quantify the variation in body composition (auxology and biphotonic absorptiometry) at the end of the randomized study (month 4) and at the end of study (month 14)
To evaluate the tolerance and safety of rhGH at the end of the randomized study (month 4) and at the end of study (month 14.

CONTACTS AND LOCATIONS:
Overall Officials: Alain LACHAUX, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Alain LACHAUX, Lyon, France